CLINICAL TRIAL: NCT01701466
Title: A Phase II Study Designed to Evaluate the Value of Neoviderm Skin Emulsion in the Prevention of Radiation Dermatitis for Patients Undergoing External Radiation Therapy
Brief Title: Neoviderm Skin Emulsion in the Prevention of Radiation Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Avario Healthcare Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Te Vuong, Director Radiation-oncology department, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-053; NCT01470872 (obsolete NCT alias)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Head and Neck Cancer; Breast Cancer
Keywords: Patients; with
MeSH Terms: conditions — Head and Neck Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm B: standard of care plus NeoVIDERM cream (Experimental): Patients will apply NeoVIDERM cream to the treatment area everyday one week before starting radiotherapy, throughout treatment and for two weeks post treatment. Patients will also perform standard of care skin treatment.
  Interventions: Other: Aveeno cream; Other: Flamazine cream; Other: NeoVIDERM cream
- Arm A: standard skin care (Active Comparator): Patients will be asked to apply Aveeno cream twice a day starting the day of their treatment until two weeks after the end of their treatments. If they develop dry desquamation, they will be asked to apply Flamazine twice a day until dermatitis resolves.
  Interventions: Other: Aveeno cream; Other: Flamazine cream

INTERVENTIONS:
Other: Aveeno cream — Twice a day
Other: Flamazine cream — Twice a day, when there is dry desquamation
Other: NeoVIDERM cream — Three times a day
  Arms: Arm B: standard of care plus NeoVIDERM cream

SUMMARY:
The purpose of this study is to determine whether NeoVIDERM is effective at preventing radiation dermatitis in patients receiving external beam radiation therapy to the head and neck or breast areas.

ELIGIBILITY:
Inclusion criteria: For patients receiving radiation to the breast

1. Patients receiving a dose of at least 50 Gy in 25 fractions with concomitant chemotherapy or treated with the McGill technique.
2. Patients able to understand and sign an informed consent form.
3. Patients that do not have active connective tissue disorders.
4. Patients 18 years or older.
5. Patients that did not receive any previous radiation.
6. Patients that do not have any known allergy to any ingredients of the NeoVIDERM cream
7. Patients need to be able to apply the creams themselves or have help with applying the creams.

Inclusion criteria: For patients receiving radiation to the head and neck

1. Patients receiving radiotherapy on fields that include both sides of the neck
2. Patients able to understand and sign an informed consent form.
3. Patients that do not have active connective tissue disorders.
4. Patients 18 years or older.
5. Patients that did not receive any previous radiation.
6. Patients that do not have any known allergy to any ingredients of the NeoVIDERM cream
7. Patients need to be able to apply the creams themselves or have help with applying the creams.

Exclusion criteria: For patients receiving radiation to the breast or the head and neck

1. Patients that have a type V or type VI skin type according to the Fitzpatrick scale (because these patients will likely have less radiodermatitis and if they do, it will be harder to evaluate it).

   The Fitzpatrick Scale:
   * Type I (scores 0-7) White; very fair; freckles. Always burns, never tans
   * Type II (scores 8-16) White; fair. Usually burns, tans with difficulty
   * Type III (scores 17-25) Beige; very common. Sometimes mild burn, gradually tans
   * Type IV (scores 25-30) Beige with a brown tint; typical Mediterranean Caucasian skin.

   Rarely burns, tans with ease
   * Type V (scores over 30) Dark brown. Very rarely burns, tans very easily
   * Type VI Black. Never burns, tans very easily
2. Allergic to any ingredient in Neoviderm cream

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum skin toxicity | 7 weeks post beginning of radiation treatments
  The objective of this study is to determine the occurrence and degree of acute skin toxicity in patients receiving radical radiation therapy with preventive application of neoVIDERM compared to patients treated with institutional standard skin care.

CONTACTS AND LOCATIONS:
Overall Officials: Te Vuong, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada